CLINICAL TRIAL: NCT00561236
Title: Low Dose (1mcg ) ACTH Stimulation Test for Assessment of the Hypothalamo- Pituitary- Adrenal Axis in Patients Treated With Intravitreal Injection of Triamcinolone Acetonide
Brief Title: Does Intravitreal Injection of Triamcinolone Acetonide Impairs the Adrenal Function
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, avraham ishay, Dr, HaEmek Medical Center, Israel
Other Study IDs: 002507EMC
Record Dates: First submitted 2007-11-18; First posted 2007-11-20 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Secondary Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The use of intravitreal corticosteroids in the management ocular inflammatory diseases has recently gained widespread acceptance. The purpose of this study is to determine if the use of intravitreal triamcinolone is associated with suppression of endogenous cortisol production, as generally admitted for patients treated with oral or parenteral corticosteroid therapy.

DETAILED DESCRIPTION:
The normalcy of hypothalamic- pituitary- adrenal axis (HPA axis) of enrolled subjects will will be assessed before intravitreal injection of 4mg of triamcinolone and again after one day, one week and two weeks. Patients with abnormal HPA axis will be re-tested after four weeks and later until the HPA axis function return to normal. The HPA axis will be assessed with low dose (1mcg) intravenous corticotropin(ACTH) stimulation test, in which cortisol levels will be sampled before , 30 minutes and 60 minutes after 1mcg ACTH IV injection.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving intravitreous injection of triamcinolone 4mg

Exclusion Criteria:

* patients receiving steroids in any form, except by intravitreous administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital-based ophtalmologic clinic
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Ishay, MD, Principal Investigator — Haemek Medical Center , Endocrine Institute
Locations (1):
- Haemek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No